CLINICAL TRIAL: NCT05358171
Title: Ultra-processed Food Consumption, Gut Microbiota, and Glucose Homeostasis in Mid-life Adults
Brief Title: Ultra-processed Food Consumption, Gut Microbiota, and Glucose Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Brenda Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-974
Record Dates: First submitted 2022-04-22; First posted 2022-05-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Insulin Sensitivity; 24-hour Glucose Control
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIgh UPF (Ultra-processed foods) (Experimental): Participants will consume a diet containing 81% total energy from UPF for 6 weeks
  Interventions: Other: HIgh UPF controlled diet
- No UPF (Active Comparator): Participants will consume a diet containing 0% total energy from UPF for 6 weeks
  Interventions: Other: No UPF controlled diet

INTERVENTIONS:
Other: HIgh UPF controlled diet — Following a two- week eucaloric lead-in diet, participants will be provided and consume a diet emphasizing UPF (81% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, pre- and probiotics, and overall diet quality, for 6 weeks.
  Arms: HIgh UPF (Ultra-processed foods)
Other: No UPF controlled diet — Following a two- week eucaloric lead-in diet, participants will be provided and consume a diet without UPF (0% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, pre- and probiotics, and overall diet quality, for 6 weeks.
  Arms: No UPF

SUMMARY:
Advancing age is associated with gut dysbiosis, low-grade chronic inflammation, progressive insulin resistance, and increased risk of type 2 diabetes (T2D). Prediabetes is present in 45-50% of middle-aged/older adults, and declines in glucose tolerance are evident in the third or fourth decade of life. Thus, there is an urgent need to identify new approaches for the prevention of type 2 diabetes among middle-aged adults. Observational research has linked intake of ultra-processed foods (UPF), which comprise ~60% of total energy intake in US adults, with increased risk of T2D. Ex vivo and animal research suggests that components of UPF alter gut microbiota composition and initiate a cascade of events leading to intestinal inflammation and impaired glycemic control. Whether mid-life adults (aged 45-65 yrs) are susceptible to the adverse impact of UPF consumption on glucose homeostasis is unknown. The overall objective of this study is to establish proof-of-concept for an impairment in glucose homeostasis following increases in UPF consumption in mid-life adults, in order to conduct a larger, more comprehensive and mechanistic trial in the future. In addition, changes in gut microbial composition and function, intestinal inflammation and permeability, serum endotoxin concentrations, and inflammatory cytokines as potential mechanisms by which UPF consumption influences glucose homeostasis will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Weight stable for previous 6 months
* Sedentary to recreationally active
* No plans to gain/lose weight or change physical activity level
* Willing to pick up food daily and consume foods provided for an 8-week period
* Verbal and written informed consent
* Approval by Medical Director
* Estrogen or testosterone usage is acceptable, if on stable dose for >6 months

Exclusion Criteria:

* BMI >35 kg/m2
* Diabetes or diabetes medication
* Antibiotic, prebiotic or prebiotic use in prior 3 months
* TCHOL >6.2 mmol/L; TG >4.5 mmol/L
* Blood pressure (BP) > 159/99 mmHg (Stable BP on antihypertensive medications used for >6 months is acceptable)
* Diagnosed inflammatory bowel disease
* Past or current heart diseases, stroke, respiratory disease, endocrine or metabolic disease, or hematological-oncological disease
* Vegetarian or vegan
* Pregnant or plans to become pregnant
* Food allergies or aversions
* 3 or fewer stools per week or regular laxative use

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity from baseline to 6-weeks post high or no UPF diet | 2 timepoints (standardized diet lead-in [baseline]), 6-weeks post high or no UPF diet, 2-hour test in laboratory
  Insulin sensitivity assessed using a 2-hour oral glucose tolerance test (75g glucose load). Blood will be collected at baseline (fasting), and thereafter at 30-minute intervals (5 total measurements in 2 hours) at baseline and post 6-weeks high or no UPF diet.

SECONDARY OUTCOMES:
Change in 24-hour glucose control (24-hour mean) from baseline to 6-weeks post high or no UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  24-hour glucose control (24-hour mean glucose concentration) will be assessed using continuous glucose monitoring for a 6-day period at baseline and post high or no UPF diet.
Change in 24-hour glucose control (AUC) from baseline to 6-weeks post high or no UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  24-hour glucose control (24-hour AUC) will be assessed using continuous glucose monitoring for a 6-day period at baseline and post high or no UPF diet.
Change in 24-hour glucose control (time in range) from baseline to 6-weeks post high or no UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  24-hour glucose control (time in range) will be assessed using continuous glucose monitoring for a 6-day period at baseline and post high or no UPF diet.
Change in 24-hour glucose control (glycemic variability [GV]) from baseline to 6-weeks post high or no UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  24-hour glucose control (GV) will be assessed using continuous glucose monitoring for a 6-day period at baseline and post high or no UPF diet.
Change in 24-hour glucose control (postprandial glucose) from baseline to 6-weeks post high or no UPF diet | 6-day measurement during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Free-living postprandial glucose concentration will be assessed using continuous glucose monitoring for a 6-day period at baseline and post high or no UPF diet.
Change in inflammatory cytokines from baseline to post 6-weeks high or no UPF diet | 5-minute blood collection in the laboratory, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Inflammatory Cytokines, including TNF alpha, IL-6, and MCP-1 will be measured by ELISA (American Diagnostica Inc).
Change in endotoxin from baseline to post 6-weeks high or no UPF diet | 5-minute blood collection in the laboratory, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Serum endotoxin will be assessed using the PyroGene Recombinant Factor C endotoxin assay (Lonza, Basel, Switzerland).
Change in gut microbial composition from baseline to post 6-weeks high or no UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Stool samples will be collected daily for 3 days before and during the final 3 days of the diet interventions. Samples will be collected daily and placed in sterile plastic containers, stored in personal freezers, and placed in coolers for transport then immediately frozen at -80°C until final processing and analysis.
Change in gut microbial function from baseline to post 6-weeks high or no UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Stool samples will be collected daily for 3 days before and during the final 3 days of the diet interventions. Samples will be collected daily and placed in sterile plastic containers, stored in personal freezers, and placed in coolers for transport then immediately frozen at -80°C until final processing and analysis.
Change in intestinal inflammation from baseline to post 6-weeks high or no UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Intestinal inflammation will be assessed using fecal calprotectin, lactoferrin, and lipocalin-2, measured using ELISA.
Change in intestinal permeability from baseline to post 6-weeks high or no UPF diet | 3-day collection during free-living, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Intestinal permeability will be assessed using serum zonulin (Immunodiagnostik AG, Bensheim, Germany) concentrations, measured using ELISA.

OTHER OUTCOMES:
Change in brachial artery function from baseline to 6-weeks post high or no UPF diet | 30-minute measurement in the laboratory, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Flow Mediated Dilation of the brachial artery will be assessed using duplex ultrasonography (GE Logiq e) with a high resolution linear array transducer. Reactive hyperemia will be produced by inflation of a pediatric BP cuff around the forearm for 5 minutes. Off line analysis of baseline and post-reactive hyperemic diameters and velocities will be performed using edge detection software (Vascular Analysis Tools, Medical Imaging Applications, Inc). Endothelium independent vasodilation (EID) will be assessed by measuring brachial arterial dilation for 10 minutes following administration of 0.4 mg of sublingual nitroglycerine. Both FMD and EID will be expressed as mm and % change from baseline diameter.
Change in arterial stiffness (Carotid femoral pulse wave velocity) from baseline to 6-weeks post high or no UPF diet | 45-minute measurement in the laboratory, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Carotid femoral (C-F) pulse wave velocity (PWV), the primary measure of arterial stiffness, will be measured. C-F waveforms will be obtained via tonometry (NIHem, Cardiovascular Engineering, Inc). Aortic PWV will be calculated from signal averaged waveforms using the ECG as the fiducial point, and body surface measurements.
Change in arterial stiffness (Beta-stiffness index) from baseline to 6-weeks post high or no UPF diet | 45-minute measurement in the laboratory, 2 timepoints (baseline, 6 weeks post high or no UPF diet)
  Beta-stiffness index will be measured using high resolution ultrasonography and tonometry of the carotid artery.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Davy, PhD RDN, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capra BT, Hudson S, Helder M, Laskaridou E, Johnson AL, Gilmore C, Marinik E, Hedrick VE, Savla J, David LA, Davy KP, Davy BM. Ultra-processed food intake, gut microbiome, and glucose homeostasis in mid-life adults: Background, design, and methods of a controlled feeding trial. Contemp Clin Trials. 2024 Feb;137:107427. doi: 10.1016/j.cct.2024.107427. Epub 2024 Jan 4. PMID 38184104